CLINICAL TRIAL: NCT01803646
Title: Efficacy and Safety of AM-101 in the Treatment of Acute Peripheral Tinnitus 2
Brief Title: AM-101 in the Treatment of Acute Tinnitus 2
Acronym: TACTT2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Auris Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AM-101-CL-12-01
Record Dates: First submitted 2013-03-01; First posted 2013-03-04 (Estimated); Results first posted 2018-05-29 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — PDCD5 protein, rat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AM-101 injection (Experimental): AM-101
  Interventions: Drug: AM-101
- Placebo injection (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AM-101 — AM-101 gel for intratympanic injection
  Arms: AM-101 injection
Drug: Placebo — Placebo gel for intratympanic injection
  Arms: Placebo injection

SUMMARY:
The purpose of this research study is to test the safety and effectiveness of the study drug, AM-101. AM-101 is tested for the treatment of tinnitus that started as the result of an injury to the inner ear or due to middle ear inflammation (otitis media). Subjects with tinnitus can take part in the study, if their tinnitus started within the last 3 months.

DETAILED DESCRIPTION:
This phase III study is assessing the drug's safety and is aiming to demonstrate efficacy of repeated intratymanic AM-101 injections in the treatment of acute peripheral tinnitus (up to 3 months from onset).

ELIGIBILITY:
Inclusion Criteria:

1. Persistent subjective peripheral tinnitus (unilateral or bilateral) following traumatic cochlear injury (acute acoustic trauma, blast trauma, middle ear surgery, inner ear barotrauma, tympanic membrane trauma) or otitis media with onset no longer than 3 months prior to randomization
2. Age ≥ 18 years and ≤ 75 years (≥ 14 years and ≤ 75 years at selected sites);
3. Negative pregnancy test (woman of childbearing potential);
4. Willing and able to use adequate hearing protection, respectively to refrain from engaging in activities or work involving loud noise exposure where sufficient hearing protection is not possible or ensured;
5. Willing and able to protect ear canal and middle ear from water exposure as long as tympanic membrane is not fully closed.

Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

1. Fluctuating tinnitus;
2. Intermittent tinnitus;
3. Tinnitus resulting from traumatic head or neck injury;
4. Presence of chronic tinnitus;
5. Meniere's Disease, history of endolymphatic hydrops, or history of fluctuating hearing loss;
6. History of repeated idiopathic sudden sensorineural hearing loss or history of acoustic neuroma;
7. Ongoing acute or chronic otitis media or otitis externa;
8. Other treatment of tinnitus for the study duration;
9. Known hypersensitivity, allergy or intolerance to the study medication or any history of severe, abnormal drug reaction;
10. Women who are breast-feeding, pregnant or who are planning to become pregnant during the study;
11. Women of childbearing potential who are unwilling or unable to practice contraception, such as hormonal contraceptives, double barrier, sexual abstinence or intercourse with a partner who has been vasectomised for at least three months;
12. Concurrent participation in another clinical study or participation in another clinical study within 30 days prior to randomization.

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2014-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medpace, Cincinnati, Ohio, United States

REFERENCES:
- [Result] Staecker H, Morelock M, Kramer T, Chrbolka P, Ahn JH, Meyer T. Safety of Repeated-Dose Intratympanic Injections with AM-101 in Acute Inner Ear Tinnitus. Otolaryngol Head Neck Surg. 2017 Sep;157(3):478-487. doi: 10.1177/0194599817711378. Epub 2017 Jun 13. PMID 28608739

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 86 sites were initiated in Canada, the United States, the Czech Republic, Israel, Turkey and Republic of South Korea. In total, 69 sites screened each at least 1 subject and 64 sites randomized subjects for treatment.
Pre-assignment Details: A total of 478 subjects were screened, 343 subjects were randomized, and 336 subjects were treated. 7 subjects were randomized (3 to AM-101 and 4 to placebo) but not treated; these subjects were excluded from the analysis sets.
  The majority (92%) of subjects completed the study.
Groups:
- AM-101 0.87 mg/mL Gel: Three intratympanic administration of AM-101 0.87 mg/mL gel within 5 days (D0-D4)
- Placebo Gel: Three intratympanic administration of placebo gel within 5 days (D0-D4).
Period: Overall Study
Arm/Group | AM-101 0.87 mg/mL Gel | Placebo Gel
Started | 204 | 139
Completed | 187 | 129
Not Completed | 17 | 10
Not completed — Protocol Violation | 1 | 0
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 9 | 6
Not completed — Randomization error | 1 | 2
Not completed — Lost to Follow-up | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AM-101 0.87 mg/mL Gel | Placebo Gel | Total
Number analyzed (Participants) | 204 | 139 | 343
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 188 | 125 | 313
  >=65 years | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (14.6) | 44.2 (15.2) | 43.7 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 37 | 80
  Male | 161 | 102 | 263
Region of Enrollment [Number; unit: participants]
  United States | 122 | 82 | 204
  Czechia | 38 | 26 | 64
  Canada | 20 | 14 | 34
  Israel | 2 | 1 | 3
  South Korea | 15 | 12 | 27
  Turkey | 7 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Change in Patient-reported Tinnitus Loudness Questionnaire (TLQ) Improvement From Baseline to Follow up Visit 3 (FUV3)
Description: Starting at the screening visit (SV), each subject recorded the following numerical rating scales (NRS) throughout the entire study duration:
  - Tinnitus loudness "at its loudest" within the last 24 hours (Tinnitus Loudness Questionnaire [TLQ] NRSLoudest). Subjects were asked "On a scale from 0 to 10, where 0 represents no tinnitus and 10 represents extremely loud tinnitus, what one number best describes your tinnitus at its loudest in the last 24 hours (including right now)?" TLQ NRSLoudest was collected from SV (D-14) to the evening before FUV3 (D83). The ratings were to be recorded every day before going to sleep on an electronic device.
  As Baseline the10 ratings of the screening period before the first treatment were averaged. For the FUV3 endpoint, the ratings of the 7 days before FUV3 were averaged.
Time Frame: Screening (D-14) versus final follow-up (D83)
Population: Valid for Efficacy dataset includes all subjects treated with at least one i.t. injection (AM-101 or placebo), a valid TLQ NRSLoudest or TFI rating at baseline and at least one valid post-baseline rating.
  Ten subjects had neither TLQ nor TFI baseline and 2 subjects had no valid rating for the TLQ resulting in 324 evaluable subjects.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | AM-101 0.87 mg/mL Gel | Placebo Gel
Number analyzed (Participants) | 195 | 129
units on a scale | 0.80 [0.51 to 1.08] | 0.63 [0.38 to 0.87]
Statistical Analysis 1: Comparison: AM-101 0.87 mg/mL Gel vs Placebo Gel; Test type: Superiority; p = 0.32, Mixed Models Analysis; Mean Difference (Net) = -0.17, 95% CI 2-sided [-0.51 to 0.17]

2. Primary Outcome: Co-Primary Efficacy: Improvement in Tinnitus Functional Index (TFI) Total Score From Baseline to FUV3
Description: The TFI was recorded on an electronic device (electronic patient reported outcome) at Treatment Visit 1 (TV1), before randomization, and at Follow up Visit 1 (FUV1), FUV2 and FUV3.
  The TFI is a patient reported outcome questionnaire and contains 25 questions. It includes eight subscales: Intrusive, Sense of Control, Cognitive, Sleep, Auditory, Relaxation, Quality of Life, and Emotional. Each question is to be rated on a NRS between 0 and 10 (or 0 to 100%), with a recall period of "over the past week".
  The TFI total score is considered as valid if there are evaluable answers for at least 19 of the 25 items (76% of items) (Meikle et al. 2012). The repondent's overall TFI score is within a 0-100 range. For the subscales the range is the same. A lower value represents an improvement for all scales.
  Please refer to the following publicly available link for more information: http://download.lww.com/wolterskluwer_vitalstream_com/PermaLink/EANDH/A/EANDH_2011_09_27_HENRY_200593_SDC15.pdf
Time Frame: D0 (=TV1) versus Day 84 (=FUV3)
Population: Valid for Efficacy dataset includes all subjects treated with at least one i.t. injection (AM-101 or placebo), a valid TLQ NRSLoudest or TFI rating at baseline and at least one valid post-baseline rating.
  Ten subjects had neither TLQ nor TFI baseline plus additional 25 subjects had no baseline for the TFI resulting in 301 evaluable subjects.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | AM-101 0.87 mg/mL Gel | Placebo Gel
Number analyzed (Participants) | 180 | 121
units on a scale | 10.4 [6.5 to 14.3] | 9.6 [5.9 to 13.3]
Statistical Analysis 1: Comparison: AM-101 0.87 mg/mL Gel vs Placebo Gel; Test type: Superiority; p = 0.63, Mixed Models Analysis; Mean Difference (Net) = -0.79, 95% CI 2-sided [-4 to 2.4]

3. Primary Outcome: Safety: Frequency of Subjects With Deterioration of Hearing at Follow up Visit 2 (FUV2)
Description: Occurence of deterioration of hearing (Air and Bone conduction) in the treated ear at FUV2.
  Deterioration is defined as a deterioration of hearing threshold of at least 15 dB from Baseline at the average of 2 contiguous frequencies.
Time Frame: Day 35
Population: Valid for Safety dataset was used. Of the 336 valid for safety subjects, 323 could be evaluated for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | AM-101 0.87 mg/mL Gel | Placebo Gel
Number analyzed (Participants) | 193 | 130
Participants
  Air conduction: Subjects with hearing deterioration | 12 | 9
  Air conduction: Subjects without hearing deterioration | 181 | 121
  Bone conduction: Subjects with hearing deterioration | 3 | 4
  Bone conduction: Subjects without hearing deterioration | 190 | 126
Statistical Analysis 1: Comparison: AM-101 0.87 mg/mL Gel vs Placebo Gel; Analysis for air conduction; Test type: Superiority; p = 0.821, Fisher Exact
Statistical Analysis 2: Comparison: AM-101 0.87 mg/mL Gel vs Placebo Gel; Analysis for bone conduction; Test type: Superiority; p = 1.0, Fisher Exact

ADVERSE EVENTS:
Time Frame: Assessed by Investigator at all Visits from Screening Visit (SV, D-14) to end of treatment visit FUV3 (D84). Including at treatment visit 1 (TV1), TV2, TV3, FUV1 and FUV2. It was also assessed at Conditional Visits if they were required.
Description: Safety population includes 336 instead of 343 subjects. As 7 subjects were randomized but not treated (see pre-assignment details).
Arm/Group | AM-101 0.87 mg/mL Gel | Placebo Gel
All-Cause Mortality (participants affected / at risk) | 0/201 | 0/135
Serious Adverse Events (participants affected / at risk) | 5/201 | 1/135
Other Adverse Events (participants affected / at risk) | 63/201 | 38/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AM-101 0.87 mg/mL Gel (N=201) | Placebo Gel (N=135)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Mental disorder (Psychiatric disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AM-101 0.87 mg/mL Gel (N=201) | Placebo Gel (N=135)
Dizziness (Nervous system disorders) | 10 | 1
Headache (Nervous system disorders) | 11 | 6
Injection site pain (General disorders) | 5 | 1
Ear discomfort (Ear and labyrinth disorders) | 14 | 8
Ear pain (Ear and labyrinth disorders) | 16 | 10
Hypoacusis (Ear and labyrinth disorders) | 8 | 4
Tinnitus (Ear and labyrinth disorders) | 8 | 5
Tympanic membrane perforation (Ear and labyrinth disorders) | 5 | 4
Vertigo (Ear and labyrinth disorders) | 2 | 4
Anxiety (Psychiatric disorders) | 7 | 1
Insomnia (Psychiatric disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 4 | 2
Nasopharyngitis (Infections and infestations) | 6 | 4
Sinusitis (Infections and infestations) | 4 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator agrees to submit a copy of any intended communication, presentation or publication (abstract, poster, article, etc.) (all together "Communication") at least 2 month in advance of the submission of proposed Communication. The Sponsor shall have 60 days, after receipt of said copies, to object to such proposed Communication. In case of such objection, the Investigator shall refrain from making such Communication for 6 months from date of receipt of such objection.